CLINICAL TRIAL: NCT04562428
Title: The Safety and Efficacy Evaluation of XSLJZ in Advanced Hepatocellular Carcinoma Patients With Multiple Protein Kinase Inhibitor Therapy: A Randomized, Double-Blind, Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH109-REC1-085
Record Dates: First submitted 2020-09-17; First posted 2020-09-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; multiple protein kinase inhibitor therapy; Xiang Sha Liu Jun Zi Decoction; appetite
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XSLJZ (Experimental): Xiang Sha Liu Jun Zi Decoction dry powder 7.5g/day tid
  Interventions: Drug: Xiang Sha Liu Jun Zi Decoction dry powder
- XSLJZ Placebo (Placebo Comparator): 10%Xiang Sha Liu Jun Zi Decoction dry powder 7.5g/day tid
  Interventions: Drug: XSLJZ Placebo

INTERVENTIONS:
Drug: Xiang Sha Liu Jun Zi Decoction dry powder — the principles of Chinese medicine treatment areinvigorating Pi, regulating qi, dissipating dampness and appetizing wei
  Arms: XSLJZ
Drug: XSLJZ Placebo — XSLJZ Placebo
  Arms: XSLJZ Placebo

SUMMARY:
The purpose of the study was search the safety and efficacy of the of Xiang Sha Liu Jun Zi Decoction (XSLJZ) in advanced hepatocellular carcinoma patients with multiple protein kinase inhibitor therapy. Evaluate the treatment effect on the symptoms of appetite and quality of life in advanced hepatocellular carcinoma patients

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the top fourth most common cancer in Taiwan. Approximately 85% of cases of HCC patients had chronic HBV or HCV infection in Taiwan. Metabolic risk factors, such as obesity, fatty liver, high lipidemia, and diabetes mellitus are associated with increased risk for nonviral hepatocellular carcinoma.

The first and second-line systemic therapy approved in advanced hepatocellular carcinoma are multikinase inhubitors .Sorafenib (Nexavar)、Regorafenib and Lenvatinib are significantly improve survival in patients who had unresectable advanced and/or metastatic HCC not amenable to local treatment methods. General fatigue, poor appetite and pain are regarded as common and unavoidable side effect experienced during the course of cancer and its treatment. Anorexia is a common cause of malnutrition and is associated with negative effects on the quality of life (QOL) for patients with cancer. However, quality of life as a prognostic factor for survival in hepatocellular carcinoma. Management of appetite is the key to improving both the QOL and the prognosis for such patients.

Cancer-related anorexia and target therapy-induced anorexia is very important in HCC patients. According to Chinese medicine theory., "spleen-deficiency, qi-stagnation and dampness" are the most common syndrome in advanced hepatocellular carcinoma patients. Thus, the principles of Chinese medicine treatment are invigorating Pi, regulating qi, dissipating dampness and appetizing wei. Most patients received traditional Chinese medicine treatment as adjuvant therapy to alleviate cancer symptoms, diminishing the side effects and complications of treatment course at late stages. The purpose of the study was search the safety and efficacy of the of Xiang Sha Liu Jun Zi Decoction (XSLJZ) in advanced hepatocellular carcinoma patients with multiple protein kinase inhibitor therapy. Evaluate the treatment effect on the symptoms of appetite and quality of life in advanced hepatocellular carcinoma patients

ELIGIBILITY:
Inclusion Criteria:

1. Advanced hepatocellular carcinoma patient
2. use multiple protein kinase inhibitor therapy paid by National Health Care Insurance system (NHCIS) in Taiwan
3. Child-Pugh A class
4. Eastern Cooperative Oncology Group performance status of 0-2
5. survival period over 3 months
6. used Xiang Sha Liu Jun Zi Decoction for one month before the multiple protein kinase inhibitor therapystarting point

Exclusion Criteria:

1. combine other cancer at the same time
2. ESRD under dialysis
3. heart disease,CHF、CAD、arrhythmia、hypertension (SBP>150mmHg，DSP>90 mmHg)
4. current serious infection
5. GI bleeding within 30 days
6. receive organ transplant
7. Child-Pugh Class B or C liver status。
8. Refractory Ascites in Liver Cirrhosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
body weight | 8 weeks
  patient body weight
EORTC QLQ-C30 score | 8 weeks
  European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire score
EORTC QLQ-HCC18 | 8 weeks
  European Organization for Research and Treatment of Hepatocellular carcinoma Core Quality of Life Questionnaire score
CASQ | 8 weeks
  cancer appetite and symptom questionnaire
FACT-G | 8 weeks
  Functional Assessment of Cancer Therapy - General

SECONDARY OUTCOMES:
CCMQ | 8 weeks
  Chinese medicine questionnaire
tong diagnosis | 8 weeks
  tong diagnosis by Automatic Tongue Diagnosis System
pulse diagnosis | 8 weeks
  pulse diagnosis by Huang's Sphygmography in Frequeny-domained Parameters

CONTACTS AND LOCATIONS:
Overall Officials: YuanChing Liao, Principal Investigator — China Medial University
Locations (1):
- China Medical University hospital, Taichung, 西屯區, Taiwan